CLINICAL TRIAL: NCT07191340
Title: A Prospective, Randomized, Single-Blinded, Crossover Clinical Trial Evaluating the Use of Noninvasive Transcutaneous Vagal Nerve Stimulation (tcVNS) for Neuromodulating the Conscious State
Brief Title: Noninvasive Transcutaneous Vagal Nerve Stimulation (tcVNS) for Neuromodulating the Conscious State
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Withdrew study equipment issue.
Sponsor: Northwestern University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STU00217188
Record Dates: First submitted 2024-03-22; First posted 2025-09-24 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Anesthesia; Delirium; Depression; Cognitive Function
Keywords: Vagal Nerve Stimulator; Post Anesthesia Care; Post Surgical
MeSH Terms: conditions — Delirium; Depression

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Participant, Outcomes Assessor
Masking Description: Participant and outcomes assessor will not know which treatment arm the subject has been assigned to during the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Treatment Group Stimulation of Vagus Nerve (Active Comparator): Stimulation of the vagus nerve with nerve stimulator placed on neck
  Interventions: Device: Vagus nerve stimulator
- Sham Placebo Group No Stimulation to Vagus Nerve (Placebo Comparator): Nerve stimulator placed on neck but not activated.
  Interventions: Device: Placebo comparator sham

INTERVENTIONS:
Device: Vagus nerve stimulator — Vagus nerve stimulator placed on neck and activated
  Arms: Treatment Group Stimulation of Vagus Nerve
Device: Placebo comparator sham — Vagus nerve stimulator placed on neck and not activated
  Arms: Sham Placebo Group No Stimulation to Vagus Nerve

SUMMARY:
The purpose of this study is to examine whether noninvasive, transcutaneous vagal nerve stimulation (tcVNS) (Gammacore Sapphire Device) can help restore consciousness in patients in the Operating Room and Post Anesthesia Care Unit (PACU). To examine whether tcVNS administered in the PACU can help reduce delirium and depression post-surgery, speeding up cognitive recovery from anesthesia, and finally determine if tcVNS can expedite discharge from the PACU.

ELIGIBILITY:
Inclusion Criteria:

* Aged > 18 years of age
* Patients undergoing lumbar surgery for degenerative disc disease or spinal stenosis involving two or more levels
* Mini-Mental State Examination (MMSE) score ≥ 15-accept mild
* Ability to use a keyboard
* Able to understand and communicate in English
* Be able to consent independently
* Women of child-bearing age must be comfortable confirming a negative pregnancy prior to participating in the study.
* Must not be involved in any other research intervention study testing neurobehavioral functioning
* Good internet connectivity and ability to use computer, smart phone or good telephone connectivity (follow up)

Exclusion Criteria:

* Age < 18 years of age
* History of vagotomy (cutting the vagus nerve)
* History of bradycardia, heart block, prolonged QT syndrome, brugada syndrome, heart failure with ejection fraction less than 35% and/or New York Heart Association symptoms
* MMSE < 15
* History of seizure disorder or intracranial hemorrhage
* Patients with carotid stenosis
* Patients with aneurysms
* Other neurological diagnoses or a diagnosis of severe psychiatric disorder (e.g., psychosis) or a reported childhood learning disability
* Pregnancy, breastfeeding
* Active addiction history
* ECG adhesive allergy
* Severe aphasia, preventing subject from understanding the protocol and giving written consent
* Patients with an active implantable medical device, such as a pacemaker, hearing aid implant, or any implanted electronic device
* Patients with metallic device such as a stent, bone plate or bone screw implanted at or near their neck
* Patients with an active implantable medical device, such as a pacemaker, hearing aid implant, or any implanted electronic device
* Patients with metallic device such as a stent, bone plate or bone screw implanted at or near their neck
* Patients who are using another device at the same time (e.g., transcutaneous electrical nerve stimulation (TENS) Unit, muscle stimulator) or any portable electronic device (e.g., mobile phone).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-10 (Estimated); Primary Completion 2023-10 (Estimated); Study Completion 2023-11 (Estimated)

PRIMARY OUTCOMES:
Aim 1: To determine if administering tcVNS enhances recovery from anesthesia | 60 minutes
  Time to a Patient State Index™ (PSi, Sedline Sedation Monitor, Massimo, Inc, Irvine, CA) score of 85.The PSi is a quantitative score derived from 4 channel EEG monitoring of the frontal and prefrontal cortex for assessing level of consciousness during sedation and general anesthesia. The score ranges from 0 (EEG suppression) to 100 (fully awake). A PSi range of 25-50 indicates optimal hypnotic state for general anesthesia.
To determine if administering tcVNS improves Richmond Agitation-Sedation Scale (RASS) scores after anesthesia | 60 minutes
  RASS Score on arrival to the PACU then 10, 15, 30, 45 and 60 min later.The Richmond Agitation-Sedation Scale (RASS) is a standardized instrument to assess arousal, cognition, and sustainability to stepped progression of stimuli. The patient is first observed. If alert a score between 1 to 4 is assigned based on their cognitive state. If the patient is not alert, the patient's name is loudly spoken and they are instructed to open their eyes and look at the speaker. This is repeated once if necessary. If there is eye opening and eye contact for > 10 seconds, a score of -1 is assigned. If not sustained for 10 secs then a score of -2 is assigned, and so forth.

SECONDARY OUTCOMES:
To determine if tcVNS can improve conscious cognitive control in post-surgical patients. | 1 month after surgery
  Targeted tcVNS compared to sham tcVNS will reduce PACU and hospital ward delirium and post-surgical depression. The investigators will test this hypothesis by PACU and in-hospital evaluations for delirium and in-hospital measurement of depression prior to discharge and at a one-month virtual follow-up evaluation.

CONTACTS AND LOCATIONS:
Overall Officials: Alyson Engle, MD, Principal Investigator — Northwestern Univesity